CLINICAL TRIAL: NCT04557293
Title: Effort-based Decision-making as a Possible Predictor of Poor Adherence to CPAP Treatment in Obstructive Sleep Apnea
Brief Title: Effort-based Decision-making and CPAP Adherence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Istituto Universitario di Studi Superiori Pavia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2425
Record Dates: First submitted 2020-08-31; First posted 2020-09-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea; Adherence
Keywords: apnoea; effort based decision making; rehabilitation; adherence
MeSH Terms: conditions — Sleep Apnea, Obstructive; Apnea | interventions — Continuous Positive Airway Pressure; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP Treatment (Experimental): Patients with OSA will undergo cognitive assessment before starting CPAP treatment and after six months of CPAP use.
  Interventions: Device: Continuous Positive Airway Pressure (CPAP) treatment
- Control Group (No Intervention): We will enrol a control group of subjects without sleep disorders and comparable to OSA patients for age and schooling. Control group will undergo cognitive assessment.

INTERVENTIONS:
Device: Continuous Positive Airway Pressure (CPAP) treatment — Treatment of Obstructive sleep apnoea syndrome with CPAP
  Arms: CPAP Treatment

SUMMARY:
Obstructive sleep apnoea is the most common sleep disorder in general population, and is often associated with cognitive deficit, mood disorders, hypertension, diabetes mellitus, excessive daytime somnolence, nicturia and an increased cardiovascular and metabolic risk. The gold standard of treatment is Continuous Positive Airway Pressure (CPAP), but the adherence is often poor. The aim of our study is to investigate the effort based-decision making in patients with OSA, pre and post CPAP treatment, as a possible cause of poor adherence.

DETAILED DESCRIPTION:
Obstructive sleep apnea is a very common disease in general population (24% males; 9% females), characterized by frequent partial or total upper-airway collapse, intermittent hypoxia, arousal from sleep, change in blood pressure, excessive daytime sleepiness, cardiovascular and metabolic diseases, psychological and cognitive consequences. The gold standard treatment is Continuous Positive Airway Pressure (CPAP), but the adherence is often poor. Poor therapy adherence might be partially explained by executive deficits, decreasing the ability to plan and pursue longsighted behaviors entailing immediate costs/efforts. We investigate the cognitive function, in particular effort based-decision making and the relationship with excessive daytime somnolence and other cognitive function in a group of OSA patients and in control group. We assess cognitive function in OSA patients at the diagnosis moment and after six months of CPAP use.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* AHI±15

Exclusion Criteria:

* BMI ≥ 35 Kg/m2
* MMSE <24
* Complex sleep apnoea
* Sleep disorder
* Psychiatric disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Memory | Change will be assesd before starting CPAP and after six months of CPAP treatment
  Short and Long-term memory will be assessed with Digit span and California verbal learning test
Executive Function | Change will be assesd before starting CPAPT and after six months of CPAP treatment
  attentional and executive functioning will be assessed with Test of Attentional Performance (TAP)
Planning | Change will be assesd before starting CPAPT and after six months of CPAP treatment
  Planning will be assessed with Tower of London
Response inhibition | Change will be assesd before starting CPAPT and after six months of CPAP treatment
  Will be assessed with Test Go-nogo
Efforth decision making | Change will be assesd before starting CPAPT and after six months of CPAP treatment
  Will be assesses with Rapid Serial Visual Presentation (RSVP)

SECONDARY OUTCOMES:
Effect of CPAP treatment on memory | After six month of CPAP use
  Administration of Digit span and California verbal Learning test
Effect of CPAP treatment on executive function | After six month of CPAP use
  Administration of Test attentional Performance
Effect of CPAP on planning | After six month of CPAP use
  Adimnistration of Tower of London Test
Effect of CPAP on Response inhibition | After six month of CPAP use
  administration of go no go Test
Effect of CPAP on effort decision making | After six month of CPAP use
  Administration of Rapid Serial Visual Presentation (RSVP) test

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Canessa, PhD, Principal Investigator — IRCCS Istituti Clinici Scientifici Maugeri - Scuola superiore IUSS Pavia
Locations (1):
- ICS Maugeri Pavia, Pavia, Italy

REFERENCES:
- [Background] Patil SP, Ayappa IA, Caples SM, Kimoff RJ, Patel SR, Harrod CG. Treatment of Adult Obstructive Sleep Apnea with Positive Airway Pressure: An American Academy of Sleep Medicine Clinical Practice Guideline. J Clin Sleep Med. 2019 Feb 15;15(2):335-343. doi: 10.5664/jcsm.7640. PMID 30736887
- [Background] Canessa N, Castronovo V, Cappa SF, Aloia MS, Marelli S, Falini A, Alemanno F, Ferini-Strambi L. Obstructive sleep apnea: brain structural changes and neurocognitive function before and after treatment. Am J Respir Crit Care Med. 2011 May 15;183(10):1419-26. doi: 10.1164/rccm.201005-0693OC. Epub 2010 Oct 29. PMID 21037021